CLINICAL TRIAL: NCT01854138
Title: Evaluating the Efficacy of the Prevena Incision Management System in Patients Undergoing Total Knee and Hip Arthroplasty
Brief Title: Evaluating Advantages of Prevena After Hip and Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, Karl Beer, Physician, ProMedica Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KCI-1333; IRB#13-033 (Other: ProMedica Institutional Review Board)
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Infection of Total Hip Joint Prosthesis
Keywords: primary knee arthroplasty; primary hip arthroplasty; negative pressure wound therapy
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Retrospectively reviewed patients who underwent Total Knee or Hip Arthroplasty and received traditional gauze dressing to cover their clean surgical wound.
- Prevena Knee/Hip (Experimental): Prospectively enrolled patients undergoing Total Knee Arthroplasty or Total Hip Arthroplasty and receiving Prevena Incision Management System on the clean surgical wound.
  Interventions: Device: Prevena Incision Management System

INTERVENTIONS:
Device: Prevena Incision Management System — Prevena Incision Management system will be applied to clean surgical wounds of patients undergoing Total Knee Arthroplasty or Total Hip Arthroplasty, immediately post-operatively. The unit will remain in place and functional for 7-8 days.
  Other Names: negative pressure wound therapy
  Arms: Prevena Knee/Hip

SUMMARY:
Determine the extent to which application of the Prevena vacuum system to clean surgical incisions immediately following surgical procedure (total hip or total knee arthroplasty) will reduce the rates of:

* readmission to hospital for surgical intervention due to wound complications
* seroma
* hematoma
* infection compared to group of patients whose wounds were covered with traditional gauze dressings.

DETAILED DESCRIPTION:
The specific aim of this research project is to determine the effect of using the Prevena vacuum system on the rate of repeat surgical procedures and surgical site complications in patients having undergone a total knee or hip arthroplasty. It is believed that negative pressure wound therapy is effective in the promotion of healing of complicated, non-healing, and infected wounds in many settings. In light of this existing evidence, the investigators believe that applying negative pressure wound therapy to clean incisions, in the orthopedic setting, before infection or complication occur may prevent complications and lower overall cost of care for patients undergoing total hip or knee arthroplasty.

The investigators' primary hypothesis is that application of the Prevena vacuum system to a clean incision in the operating room for patients who have undergone a total knee arthroplasty or hip replacement surgery will reduce the occurrence of repeat surgeries when the system remains in place and functional for seven days following its application. Prevena is the ideal system for this patient population because it is best suited for non-draining wounds; hip and knee arthroplasties result most often in non-draining wounds, which evidence suggests are less likely to become infected and cause other complications.

Secondary hypotheses to be tested in this study are that the application and use of the Prevena vacuum system in patients who have undergone a total knee arthroplasty or hip replacement surgery will reduce the occurrence of seromas, hematomas, and will also reduce the occurrence of surgical site infections when the system remains in place and functional for seven days after application. Additionally, the investigators wish to compare the level of pain experienced by patients who use the Prevena system after surgery in comparison to those whose incision sites are covered with traditional dressings. The investigators hypothesize that patients whose wounds are dressed with the Prevena system will experience less pain than patients whose wounds are dressed with traditional dressings, which may be quite bulky and carry the risk of tape trauma injury. Finally, the investigators hypothesize that because the Prevena system will prevent surgical site complications that may lead to repeat procedures, the cost of treating patients with Prevena will be lower than the total relative cost of treating the patients whose wounds are dressed with traditional dressings.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total hip or knee arthroplasty
* 18-85 years of age

Exclusion Criteria:

* Patients undergoing revision total hip or knee arthroplasty
* Allergy to silver
* Current systemic infection
* Currently being treated for malignancy
* Patients suffering from anemia or malnutrition
* Patients afflicted with jaundice
* Patients deemed to be non-compliant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beer, MD, Principal Investigator — ProMedica Health System
Locations (1):
- Wildwood Orthopaedic and Spine Hospital, Toledo, Ohio, United States

REFERENCES:
- [Derived] Redfern RE, Cameron-Ruetz C, O'Drobinak SK, Chen JT, Beer KJ. Closed Incision Negative Pressure Therapy Effects on Postoperative Infection and Surgical Site Complication After Total Hip and Knee Arthroplasty. J Arthroplasty. 2017 Nov;32(11):3333-3339. doi: 10.1016/j.arth.2017.06.019. Epub 2017 Jun 17. PMID 28705547

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were consented at time of surgery scheduling up to six months in advance of surgery.
Groups:
- Prevena Hip/Knee: Prospectively enrolled patients undergoing Total Knee Arthroplasty or Total Hip Arthroplasy and receiving Prevena Incision Management System on the clean surgical wound.
  Prevena Incision Management System: Prevena Incision Management system will be applied to clean surgical wounds of patients undergoing Total Knee Arthroplasty, immediately post-operatively. The unit will remain in place and functional for 7-8 days.
  Prevena Incision Management system will be applied to clean surgical wounds of patients undergoing Total Hip Arthroplasty, immediately post-operatively. The unit will remain in place and functional for 7-8 days.
Period: Overall Study
Arm/Group | Control | Prevena Hip/Knee
Started | 400 (historical control with waiver of authorization; no informed consent signed) | 248
Completed | 400 | 196
Not Completed | 0 | 52

BASELINE CHARACTERISTICS:
Groups:
- Prevena Hip/Knee: Prospectively enrolled patients undergoing Total Knee Arthroplasty or Total Hip Arthroplasty and receiving Prevena Incision Management System on the clean surgical wound.
  Prevena Incision Management System: Prevena Incision Management system will be applied to clean surgical wounds of patients undergoing Total Knee Arthroplasty, immediately post-operatively. The unit will remain in place and functional for 7-8 days.
  Prevena Incision Management system will be applied to clean surgical wounds of patients undergoing Total Hip Arthroplasty, immediately post-operatively. The unit will remain in place and functional for 7-8 days.
- Total: Total of all reporting groups
Arm/Group | Control | Prevena Hip/Knee | Total
Number analyzed (Participants) | 400 | 196 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.8) | 66.9 (10.2) | 66.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 129 | 345
  Male | 184 | 67 | 251

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Readmissions
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Prevena Knee/Hip
Number analyzed (Participants) | 400 | 196
Participants | 15 | 3

2. Secondary Outcome: Number of Participants With Infection
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Prevena Hip/Knee
Number analyzed (Participants) | 400 | 196
Participants | 14 | 2

3. Secondary Outcome: Number of Participants With Seroma
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Prevena Hip/Knee
Number analyzed (Participants) | 400 | 196
Participants | 2 | 0

4. Secondary Outcome: Number of Participants With Hematoma
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Prevena Hip/Knee
Number analyzed (Participants) | 400 | 196
Participants | 9 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks postoperatively
Arm/Group | Control | Prevena Hip/Knee
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/196
Other Adverse Events (participants affected / at risk) | 9/400 | 27/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=400) | Prevena Hip/Knee (N=196)
Other reactions (Skin and subcutaneous tissue disorders) | 9 (9) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No